CLINICAL TRIAL: NCT01430442
Title: Phase IIb: Double-Blind, Randomized, Placebo Controlled, Dose-ranging Trial of BMS-927711 for the Acute Treatment of Migraine
Brief Title: Dose Ranging Study of Rimegepant (BMS-927711) for the Acute Treatment of Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN170-003
Record Dates: First submitted 2011-09-07; First posted 2011-09-08 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2022-12

CONDITIONS: Migraine; Acute Treatment of Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rimegepant sulfate; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Treatment A: Rimegepant, 10 mg (Experimental): Participants received a single dose (one capsule) of rimegepant 10 milligram (mg) orally and three rimegepant placebo-matching capsules, orally, anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
  Interventions: Drug: Rimegepant; Drug: Placebo
- Treatment B: Rimegepant, 25 mg (Experimental): Participants received a single dose (one capsule) of rimegepant 25 mg orally; and three rimegepant placebo-matching capsules, orally, anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
  Interventions: Drug: Rimegepant; Drug: Placebo
- Treatment C: Rimegepant, 75 mg (Experimental): Participants received a single dose (one capsule) of rimegepant 75 mg orally; and three rimegepant placebo-matching capsules, orally, anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
  Interventions: Drug: Rimegepant; Drug: Placebo
- Treatment D: Rimegepant, 150 mg (Experimental): Participants received a single dose (one capsule) of rimegepant 150 mg orally; and three rimegepant placebo-matching capsules, orally, anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
  Interventions: Drug: Rimegepant; Drug: Placebo
- Treatment E: Rimegepant, 300 mg (Experimental): Participants received a single dose (two 150 mg capsules) of rimegepant 300 mg orally; and two rimegepant placebo-matching capsules, orally, anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
  Interventions: Drug: Rimegepant; Drug: Placebo
- Treatment F: Rimegepant, 600 mg (Experimental): Participants received a single dose (four capsules of 150 mg each) of rimegepant 600 mg orally; anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
  Interventions: Drug: Rimegepant; Drug: Placebo
- Treatment P: Rimegepant Placebo-Matching Capsules (Placebo Comparator): Participants received a single dose (4 capsules) of rimegepant placebo-matching capsules orally, anytime within 45 days of randomization once they experienced a migraine headache of moderate to severe intensity.
  Interventions: Drug: Placebo
- Treatment G: Sumatriptan 100 mg (Active Comparator): Participants received a single dose (one capsule) of rimegepant-matching sumatriptan 100 mg orally and three rimegepant matching placebo capsules orally, anytime within 45 days of randomization once they experienced a migraine headache of moderate to severe intensity.
  Interventions: Drug: Placebo; Drug: Sumatriptan

INTERVENTIONS:
Drug: Rimegepant — Rimegepant capsules
  Arms: Treatment A: Rimegepant, 10 mg; Treatment B: Rimegepant, 25 mg; Treatment C: Rimegepant, 75 mg; Treatment D: Rimegepant, 150 mg; Treatment E: Rimegepant, 300 mg; Treatment F: Rimegepant, 600 mg
Drug: Placebo — Rimegepant placebo-matching capsules
Drug: Sumatriptan — Rimegepant matching sumatriptan and Rimegepant matching placebo capsules
  Other Names: Imitrex®
  Arms: Treatment G: Sumatriptan 100 mg

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of rimegepant (BMS-927711) compared with placebo in the acute treatment of migraine as measured by Pain Freedom (headache pain intensity level reported as "no pain") at 2 hours post dose using a four point numeric rating scale (no pain, mild pain, moderate pain, severe pain) while identifying an optimal dose to support the Phase 3 clinical trials.

DETAILED DESCRIPTION:
Intervention Model: Parallel Versus Comparator + Placebo

ELIGIBILITY:
Key Inclusion Criteria:

* Patient with at least 1-year history of migraines (with or without aura) including the following:

  * Migraine attacks more than 1 year with age of onset prior to 50 years of age
  * Migraine attacks, on average, last about 4 - 72 hours if untreated
  * No more than 8 attacks of moderate to severe intensity per month within last 3 months
  * Patient must be able to distinguish migraine attacks from tension/cluster attacks and must have consistent migraine headaches of at least 2 migraine headaches attacks of moderate to severe intensity in each of the last 3 months
  * Less than 15 days of headache (migraine or non-migraine) per month in each of 3 months prior to screening
* Male and female ≥ 18 years and ≤ age 65
* No clinically significant abnormality identified on the medical or laboratory evaluation

Key Exclusion Criteria:

* Patient has a history of basilar migraine or hemiplegic migraine
* Patient does not receive migraine relief from triptan migraine treatment
* Medications that may alter the pH of the stomach (acid reducing agents), such as H-2 antagonists, Proton Pump inhibitors (PPI), antacids
* History of ergotamine or triptan intake greater than/equal 10 days per month on a regular basis for greater than 3 months
* History of non-narcotic analgesic intake on greater then/equal 15 days per month for greater than/equal 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1026 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Clinical Res. Advantage Inc/ Desert Clinical Research Llc, Tempe, Arizona
  - University Of California, San Francisco, San Francisco, California
  - California Medical Clinic For Headache, Santa Monica, California
  - Encompass Clinical Research, Spring Valley, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Radiant Research, Inc., Denver, Colorado
  - Miami Research Associates, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Compass Research, Llc, Orlando, Florida
  - Broward Research Group, Pembroke Pines, Florida
  - Comprehensive Clinical Development, Inc, St. Petersburg, Florida
  - Diamond Headache Clinic, Ltd., Chicago, Illinois
  - Milford Emergency Associates, Inc., Milford, Massachusetts
  - Medvadis Research Corporation, Watertown, Massachusetts
  - Michigan Head Pain And Neurological Institute, Ann Arbor, Michigan
  - Clinical Research Institute, Inc., Minneapolis, Minnesota
  - The Center For Pharmaceutical Research. Pc, Kansas City, Missouri
  - Clinvest/ A Division Of Banyan Group, Inc., Springfield, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Regional Clinical Research Inc., Endwell, New York
  - Central New York Clinical Research, Manlius, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Pharmquest, Greensboro, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - Pmg Research Of Winston-Salem, Winston-Salem, North Carolina
  - Community Research, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Clinical Research Of Philadelphia, Llc, Philadelphia, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina
  - Clinsearch, Llc, Chattanooga, Tennessee
  - Premier Research Group Limited, Austin, Texas
  - Futuresearch Trials Of Neurology, Austin, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - J. Lewis Research, Inc, Salt Lake City, Utah
  - The Innovative Clinical Research Center, Alexandria, Virginia
  - Tidewater Integrated Medical Research, Virginia Beach, Virginia
  - Swedish Pain And Headache Center, Seattle, Washington

REFERENCES:
- [Derived] Marcus R, Goadsby PJ, Dodick D, Stock D, Manos G, Fischer TZ. BMS-927711 for the acute treatment of migraine: a double-blind, randomized, placebo controlled, dose-ranging trial. Cephalalgia. 2014 Feb;34(2):114-25. doi: 10.1177/0333102413500727. Epub 2013 Aug 21. PMID 23965396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 41 centers in the United States. A total of 1026 participants were enrolled in the study, and 885 of these were randomized to treatment. Of the 141 participants who were not randomized, the main reason for non-randomization was participants no longer met inclusion criteria.
Pre-assignment Details: The study was divided into 3 phases: a screening/baseline phase (3-28 days), an acute treatment phase (up to 45 days during which participants were treated on 1 migraine headache of moderate to severe intensity), followed by an end-of-treatment visit within 7 days of administration of study drug.
Groups:
- Treatment G: Sumatriptan 100 mg: Participants received a single dose (one capsule) of rimegepant-matching sumatriptan 100 mg orally and three matching placebo capsules orally, anytime within 45 days of randomization once they experienced a migraine headache of moderate to severe intensity.
Period: Overall Study
Arm/Group | Treatment A: Rimegepant, 10 mg | Treatment B: Rimegepant, 25 mg | Treatment C: Rimegepant, 75 mg | Treatment D: Rimegepant, 150 mg | Treatment E: Rimegepant, 300 mg | Treatment F: Rimegepant, 600 mg | Treatment P: Rimegepant Placebo-Matching Capsules | Treatment G: Sumatriptan 100 mg
Started | 85 | 68 | 91 | 90 | 121 | 92 | 229 | 109
Completed | 72 | 62 | 86 | 86 | 112 | 84 | 210 | 100
Not Completed | 13 | 6 | 5 | 4 | 9 | 8 | 19 | 9
Not completed — Subject Withdrew Consent | 3 | 0 | 1 | 0 | 2 | 1 | 5 | 2
Not completed — Lost to Follow-up | 2 | 0 | 1 | 2 | 2 | 1 | 5 | 1
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Patient No Longer Meets Study Criteria | 7 | 6 | 3 | 2 | 5 | 5 | 9 | 6

BASELINE CHARACTERISTICS:
Population: The analysis was performed in randomized population defined as all participants who were randomized to double-blind treatment.
Groups:
- Treatment A: Rimegepant, 10 mg: Participants received a single dose (one capsule) of rimegepant 10 mg orally and three rimegepant placebo-matching capsules, orally, anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
- Treatment B: Rimegepant, 25 mg: Participants received a single dose (one capsule) of rimegepant 25 mg orally, and three rimegepant placebo-matching capsules, orally, anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
- Treatment C: Rimegepant, 75 mg: Participants received a single dose (one capsule) of rimegepant 75 mg orally, and three rimegepant placebo-matching capsules, orally, anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
- Treatment D: Rimegepant, 150 mg: Participants received a single dose (one capsule) of rimegepant 150 mg orally, and three rimegepant placebo-matching capsules, orally, anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
- Treatment F: Rimegepant, 600 mg: Participants received a single dose (four capsules of 150 mg each) of rimegepant 600 mg orally, anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
- Total: Total of all reporting groups
Arm/Group | Treatment A: Rimegepant, 10 mg | Treatment B: Rimegepant, 25 mg | Treatment C: Rimegepant, 75 mg | Treatment D: Rimegepant, 150 mg | Treatment E: Rimegepant, 300 mg | Treatment F: Rimegepant, 600 mg | Treatment P: Rimegepant Placebo-Matching Capsules | Treatment G: Sumatriptan 100 mg | Total
Number analyzed (Participants) | 85 | 68 | 91 | 90 | 121 | 92 | 229 | 109 | 885
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (10.36) | 36.5 (11.92) | 38.5 (11.87) | 39.2 (11.26) | 41.9 (11.46) | 39.3 (13.01) | 37.9 (11.36) | 40.6 (10.47) | 39.3 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 61 | 81 | 63 | 101 | 76 | 196 | 91 | 736
  Male | 18 | 7 | 10 | 27 | 20 | 16 | 33 | 18 | 149

OUTCOME MEASURES:

1. Primary Outcome: Number of Pain Free Participants (Pain Freedom) at 2 Hours Post-dose
Description: Pain freedom was defined as participants reporting a value of "none" on the four-point numeric rating scale (none=0, mild =1, moderate =2, severe =3) from baseline. Participants with baseline moderate pain or severe pain were included in the analysis.
Time Frame: Baseline, 2 hours post-dose
Population: Efficacy population - all participants who took study medication with 1 post-randomization efficacy evaluation and a corresponding baseline pain evaluation for the treated headache. Participants with mild baseline pain are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Rimegepant, 10 mg | Treatment B: Rimegepant, 25 mg | Treatment C: Rimegepant, 75 mg | Treatment D: Rimegepant, 150 mg | Treatment E: Rimegepant, 300 mg | Treatment F: Rimegepant, 600 mg | Treatment P: Rimegepant Placebo-Matching Capsules | Treatment G: Sumatriptan 100 mg
Number analyzed (Participants) | 71 | 61 | 86 | 85 | 111 | 82 | 203 | 100
Participants | 14 | 12 | 27 | 28 | 33 | 20 | 31 | 35

2. Secondary Outcome: Number of Participants With Total Migraine Freedom at 2 Hours Post Dose
Description: Total migraine freedom is defined as complete absence of migraine symptoms. A participant was positive for total migraine freedom at a particular time point if he/she reports the absence of: pain, nausea, photophobia, and phonophobia. This corresponds to reporting "none" on each of the four-point numeric rating scale (none =0, mild =1, moderate =2, severe =3) from baseline associated with these symptoms. Participants with baseline moderate pain or severe pain were included in the analysis.
Time Frame: Baseline, 2 hours post dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Rimegepant, 10 mg | Treatment B: Rimegepant, 25 mg | Treatment C: Rimegepant, 75 mg | Treatment D: Rimegepant, 150 mg | Treatment E: Rimegepant, 300 mg | Treatment F: Rimegepant, 600 mg | Treatment P: Rimegepant Placebo-Matching Capsules | Treatment G: Sumatriptan 100 mg
Number analyzed (Participants) | 71 | 61 | 86 | 85 | 111 | 82 | 203 | 100
Participants | 13 | 11 | 24 | 22 | 26 | 16 | 24 | 32

3. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Discontinuation Due to Adverse Events
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition, unfavorable and unintended sign, symptom, or disease temporally associated with the use of study drug, whether or not related to study drug. A SAE was defined as an event which was fatal or life threatening, required or prolonged hospitalization, was significantly or permanently disabling or incapacitating, constituted a congenital anomaly or a birth defect, or suspected transmission of an infectious agent, or encompassed any other clinically significant event that could jeopardize the subject or require medical or surgical intervention to prevent one of the aforementioned outcomes.
Time Frame: AEs: from first dose to end of treatment visit (up to 7 weeks); SAE: from signing of informed consent to 30 days after the last dose (up to 11 weeks).
Population: The analysis was performed on safety population, defined as all participants in the randomized population who took at least 1 capsule of study medication, as identified on the dosing record.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Rimegepant, 10 mg | Treatment B: Rimegepant, 25 mg | Treatment C: Rimegepant, 75 mg | Treatment D: Rimegepant, 150 mg | Treatment E: Rimegepant, 300 mg | Treatment F: Rimegepant, 600 mg | Treatment P: Rimegepant Placebo-Matching Capsules | Treatment G: Sumatriptan 100 mg
Number analyzed (Participants) | 72 | 62 | 86 | 86 | 112 | 84 | 209 | 100
Participants
  AEs | 15 | 10 | 18 | 12 | 18 | 14 | 29 | 17
  SAEs | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Participants discontinued due to AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Achieving Sustained Pain Freedom From 2 to 24 Hours Post Dose
Description: Participants were considered to have sustained pain freedom if all of their reported pain readings in the interval are "none" on the four point numeric rating scale (no pain=0, mild pain=1, moderate pain=2, severe pain=3). The intervals are inclusive of the endpoints. Sustained pain freedom was analyzed with a Cochran Mantel Haenszel (CMH) test for general association that compares the ED90 to placebo, and controls for baseline pain severity.
Time Frame: 2 hours to 24 hours post dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Rimegepant, 10 mg | Treatment B: Rimegepant, 25 mg | Treatment C: Rimegepant, 75 mg | Treatment D: Rimegepant, 150 mg | Treatment E: Rimegepant, 300 mg | Treatment F: Rimegepant, 600 mg | Treatment P: Rimegepant Placebo-Matching Capsules | Treatment G: Sumatriptan 100 mg
Number analyzed (Participants) | 71 | 61 | 86 | 85 | 111 | 82 | 203 | 100
Participants | 9 | 10 | 24 | 24 | 29 | 17 | 15 | 26

5. Secondary Outcome: Number of Participants Achieving Sustained Pain Freedom From 2 to 48 Hours Post Dose
Description: Participants were considered to have sustained pain freedom if all of their reported pain readings in the interval are "none" on the four point numeric rating scale (no pain=0, mild pain=1, moderate pain=2, severe pain=3). The intervals are inclusive of the endpoints. Sustained pain freedom was analyzed with a CMH test for general association that compares the ED90 to placebo, and controls for baseline pain severity.
Time Frame: 2 hours to 48 hours post dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Rimegepant, 10 mg | Treatment B: Rimegepant, 25 mg | Treatment C: Rimegepant, 75 mg | Treatment D: Rimegepant, 150 mg | Treatment E: Rimegepant, 300 mg | Treatment F: Rimegepant, 600 mg | Treatment P: Rimegepant Placebo-Matching Capsules | Treatment G: Sumatriptan 100 mg
Number analyzed (Participants) | 71 | 61 | 86 | 85 | 111 | 82 | 203 | 100
Participants | 8 | 9 | 24 | 24 | 29 | 17 | 15 | 26

ADVERSE EVENTS:
Time Frame: AEs: from first dose to end of treatment visit (up to 52 days); SAE: from signing of informed consent to 30 days after the last dose (up to 80 days)
Description: All-Cause Mortality based on randomized population. SAEs and Other AEs based on safety population, defined as all participants in the randomized population who took at least 1 capsule of study medication, as identified on the dosing record.
Groups:
- Treatment A: Rimegepant, 10 mg: Participants received a single dose (one capsule) of rimegepant 10 mg orally, and three rimegepant placebo-matching capsules, orally, anytime within 45 days of randomization, once they experienced a migraine headache of moderate to severe intensity.
Arm/Group | Treatment A: Rimegepant, 10 mg | Treatment B: Rimegepant, 25 mg | Treatment C: Rimegepant, 75 mg | Treatment D: Rimegepant, 150 mg | Treatment E: Rimegepant, 300 mg | Treatment F: Rimegepant, 600 mg | Treatment P: Rimegepant Placebo-Matching Capsules | Treatment G: Sumatriptan 100 mg
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/68 | 0/91 | 0/90 | 0/121 | 0/92 | 0/229 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/62 | 0/86 | 3/86 | 0/112 | 0/84 | 0/209 | 0/100
Other Adverse Events (participants affected / at risk) | 4/72 | 0/62 | 3/86 | 3/86 | 6/112 | 7/84 | 5/209 | 2/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: Rimegepant, 10 mg (N=72) | Treatment B: Rimegepant, 25 mg (N=62) | Treatment C: Rimegepant, 75 mg (N=86) | Treatment D: Rimegepant, 150 mg (N=86) | Treatment E: Rimegepant, 300 mg (N=112) | Treatment F: Rimegepant, 600 mg (N=84) | Treatment P: Rimegepant Placebo-Matching Capsules (N=209) | Treatment G: Sumatriptan 100 mg (N=100)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POST LUMBAR PUNCTURE SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A: Rimegepant, 10 mg (N=72) | Treatment B: Rimegepant, 25 mg (N=62) | Treatment C: Rimegepant, 75 mg (N=86) | Treatment D: Rimegepant, 150 mg (N=86) | Treatment E: Rimegepant, 300 mg (N=112) | Treatment F: Rimegepant, 600 mg (N=84) | Treatment P: Rimegepant Placebo-Matching Capsules (N=209) | Treatment G: Sumatriptan 100 mg (N=100)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 5 (5) | 7 (7) | 5 (5) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less